CLINICAL TRIAL: NCT03740139
Title: A Trial of a Police-Mental Health Linkage System for Jail Diversion and Reconnection to Care
Brief Title: The Police-Mental Health Linkage System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Michael Compton, Professor of Psychiatry, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: AAAV1672; R01MH117191 (NIH); NYSPI 7654 (Other: New York State Psychiatric Institute)
Record Dates: First submitted 2018-10-21; First posted 2018-11-14 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Mental Disorders, Severe; Schizophrenia and Related Disorders; Bipolar Disorder; Depressive Disorder
Keywords: Serious mental illnesses; Pre-arrest jail diversion; Police
MeSH Terms: conditions — Mental Disorders; Schizophrenia; Bipolar Disorder; Depressive Disorder

STUDY DESIGN:
Intervention Model Description: Participants will be randomized either to the intervention (the "Linkage System") or to no additional intervention.
Who Masked: Participant
Masking Description: Subjects will not know the arm that they are randomized to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): The Police-Mental Health Linkage System
  In the case of an encounter between law enforcement and subjects randomized to this group, the officer will receive a notice disclosing that the participant receives services in a mental health clinic and that he/she has the opportunity to call to speak with a mental health professional.
  Interventions: Other: The Police-Mental Health Linkage System
- No Intervention (No Intervention): In the case of an encounter between law enforcement and subjects randomized to this arm of the study, the officer will not receive any notice.

INTERVENTIONS:
Other: The Police-Mental Health Linkage System — When, during an encounter, the police officer decides to call the number provided in the notice, the Linkage Specialist (a licensed mental health provider from the mental health service where the subject was recruited, who has access to the clinic's EMR) can provide telephonic support to the officer.
  Arms: Intervention

SUMMARY:
The aim of this randomized, controlled trial is to study the effectiveness of a potential new form of pre-arrest jail diversion for people with serious mental illnesses: the Police-Mental Health Linkage System. In the case of an encounter with a police officer, for half of the participants, during the background check, a message will notify the officer that the subject has mental health considerations. The notice contains a phone number of a provider working at the mental health clinic where the subject is receiving services, who can provide telephonic support to the officer. For the other half of participants, the message will not appear to the officers in the case of an encounter.

DETAILED DESCRIPTION:
Fragmentation between mental health (MH) and criminal justice (CJ) systems leads to many persons with serious mental illnesses (SMI) being arrested/incarcerated when MH treatment would be more appropriate. As defined by SAMHSA, the disorders typically meeting criteria for SMI include schizophrenia, schizoaffective disorder, other psychotic disorders, major depressive disorders, and bipolar disorders. This study aims to test the effectiveness of a new police-MH linkage system. This study is a randomized, controlled trial to study the effectiveness of our new services-level intervention. Our "linkage system" piggybacks on the Georgia's criminal justice information system such that a police officer running a routine inquiry (similar to a background check) during an encounter with a consented and enrolled outpatient with a serious mental illness will receive an electronic message to call for information that might assist them. The officer can immediately call and connect to a Linkage Specialist (licensed mental health professional in the local public mental health system where the patient is or was enrolled in outpatient care), who provides brief telephonic support, information, and advice to the officer. The investigators have shown, in the recently completed NIMH-funded R34 intervention development project, that in some cases, a discretionary arrest (i.e., not obligatory, no violence involved) is replaced by informal resolution in light of the new information provided to the officer via the inquiry message and telephonic support from the Linkage Specialist. Furthermore, even more common than jail diversion, many patients involved in a police encounter were reconnected to care (after having fallen out of care and becoming symptomatic). This trial aims to determine whether or not the new linkage system is effective for reducing arrests and reducing discontinuities (gaps) in outpatient mental health care services. Partnering with our CJ partner, Georgia Bureau of Investigation (which houses Georgia's CJ databases/information system), as well as 4 public MH agencies covering 25 counties in Georgia, the investigators will conduct a randomized trial of the linkage system involving 1,600 outpatients with SMI. The investigators will test the hypotheses that patients randomized to the linkage system (as compared to those randomized to a database that does not generate the MH notice and phone number) will: (1) be less likely to be arrested, (2) have fewer arrests (both based on administrative (rap sheet) data provided by GBI), and (3) be less likely to have gaps in outpatient MH services, as evidenced by fewer absences from care of >3 months (based on data from the MH agencies' EMRs).

ELIGIBILITY:
Inclusion Criteria:

* Receiving outpatient services from DeKalb, Gateway, Pineland, or Unison Community Service Boards in Georgia
* Able to speak/read English
* Clinical diagnosis of one of the following: psychotic disorder, bipolar disorder, or major depressive disorder
* History of at least one prior arrest within the past 5 years
* Capacity to give informed consent

Exclusion Criteria:

* Enrolled in any other research project or currently enrolled in the Opening Doors to Recovery research project
* Known or suspected intellectual disability, mental retardation, or dementia
* Known or suspected autism-spectrum disorder, organic mental disorder, and/or traumatic brain injury
* Significant medical condition compromising ability to participate (e.g., short of breath, in pain)
* Has a guardian
* Received service less than 3 times in the previous year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1405 (Actual)
Dates: Start 2019-02-06 (Actual); Primary Completion 2024-04-12 (Actual); Study Completion 2024-04-12 (Actual)

PRIMARY OUTCOMES:
Lower likelihood of being arrested and lower number of arrests for participants randomized to receive the Police-MH linkage system. | 24 months of study enrollment
  Hypothesis A: Patients randomized to the linkage system will be less likely to be arrested in the 24-month study period than those not in the system, based on administrative (rap) sheet data provided by GBI.
  Hypothesis B: Patients randomized to the linkage system will have fewer arrests than controls in that 24-month period.

SECONDARY OUTCOMES:
Lower number of absences from care of >3 months for participants randomized to receive the Police-MH linkage system. | 24 months of study enrollment
  Hypothesis C: Patients randomized to the linkage system will have fewer discontinuities in MH services, as evidenced by fewer absences from care of >3 months, based on clinical encounter data from the Community Service Boards' EMR.

CONTACTS AND LOCATIONS:
Overall Officials: Michael T Compton, MD, MPH, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - DeKalb Community Service Board, Decatur, Georgia
  - Gateway Behavioral Health Services, Savannah, Georgia

IPD SHARING:
Plan to Share IPD: Yes
Data collected from this clinical trials research will be deposited into the National database for Clinical Trials Related to Mental Illness (NDCT). In order to deposit the data, we will use a consent form that allows broad data sharing within the research community. A global unique identifier (GUID) will be created for each research participant using the software that NIMH will provide. Dr. Compton and Dr. Pauselli will work with NIMH to create data dictionaries that are relevant to their research. We will share our results, positive and negative, specific to the cohorts and outcome measures studied
Time Frame: To Be Determined
Access Criteria: To Be Determined